CLINICAL TRIAL: NCT05722171
Title: Clinical Study of UTAA06 Injection in the Treatment of Relapsed/Refractory Acute
Brief Title: Clinical Study of UTAA06 Injection in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-p002-015
Record Dates: First submitted 2023-01-16; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gdT cell injection targeting B7-H3 chimeric atigen receptor (Experimental): UTAA06 injection
  Interventions: Biological: gdT cell injection targeting B7-H3 chimeric antigen receptor

INTERVENTIONS:
Biological: gdT cell injection targeting B7-H3 chimeric antigen receptor — The subjects, who sign the informed consent forms and been screened by inclusion/exclusion criteria, will be assigned into 1E8, 2E8 and 4E8 CAR-gdT groups in order of sequence. And the subjects will be administered once.
  Other Names: UTAA06 injection

SUMMARY:
This is a single-arm, open-label, dose-escalation study to explore the safety, efficacy, and cytodynamic characteristics of the drug, and to initially observe the efficacy of the drug in subjects with relapsed/refractory B7-H3-positive acute myeloid cell line leukemia.

DETAILED DESCRIPTION:
Eligible subjects will receive 1.0×10^8 CAR gdT, 2.0×10^8 CAR gdT, 4.0×10^8 CAR gdT, or additional doses may be added at the discretion of investigator and sponsor.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age≥ 18 years old, gender is not limited;
* (2) expected survival time≥ 3 months;
* (3) ECOG score 0-1 points;
* (4) Acute myeloid leukemia was clearly diagnosed during screening, and tumor cells were positive for B7-H3 expression;
* (5) Subjects with relapsed/refractory acute myeloid leukemia who have failed standard treatment or lack effective treatment methods.
* (6) Coagulation function, liver and kidney function, cardiopulmonary function meet requirements.
* (7) Be able to understand the trial and have signed the informed consent form.

Exclusion Criteria:

* (1) Malignant tumors other than acute myeloid leukemia within 5 years before screening;
* (2) Those who test positive for virus and syphilis;
* (3) Severe heart disease: including but not limited to unstable angina, myocardial infarction (within 6 months before screening), congestive heart failure (New York Heart Association [NYHA] classification≥ grade III), severe arrhythmia;
* (4) Unstable systemic diseases judged by the investigator: including but not limited to severe liver, kidney or metabolic diseases requiring drug treatment;
* (5) Active infection or uncontrollable infection requiring systemic treatment within 7 days prior to screening;
* (6) pregnant or lactating women, female subjects who planned to become pregnant within 2 years after cell reinfusion or male subjects whose partners planned to become pregnant within 2 years after their cell reinfusion;
* (7) Subjects who were receiving systemic steroid therapy within 7 days prior to the year or who were judged by the investigator to require long-term systemic steroid therapy during treatment (other than inhalation or topical use);
* (8) Have participated in other clinical studies within 1 month before screening;
* (9) There was evidence of central nervous system invasion during subject screening, such as tumor cells detected in cerebrospinal fluid or imaging showing central infiltration;
* (10) Those who have graft-versus-host response and need to use immunosuppressants;
* (11) Those with a history of epilepsy or other central nervous system diseases;
* (12) Patients with primary immunodeficiency diseases;
* (13) situations that other investigators consider unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-12-27 (Estimated); Study Completion 2024-12-27 (Estimated)

PRIMARY OUTCOMES:
Assessment of the safety after UTAA06 injection treatment (Safety) | About 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
To evaluate anti-tumor activity (overall survival) | About 2 years
  Defined as the time from start of UTAA06 UTAA06 infusion therapy to death (due to any cause)
To evaluate anti-tumor activity (duration of response) | About 2 years
  Defined as the time from the first tumor assessment of CR or PR, CR or CRi to the first assessment of disease recurrence or progression or death (due to any cause).
To evaluate anti-tumor activity (progression free survival) | About 2 years
  Defined as the time from the start of UTAA06 infusion therapy to the first disease progression or recurrence or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, Doctor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- PersonGen Anke Cellular Therapeutice Co., Ltd., Hefei, Anhui, China